CLINICAL TRIAL: NCT07289529
Title: COMPASS 65+ - Community-based Physical Activity Snacks for Healthy Aging in Overweight and Obese Aged Adults
Acronym: COMPASS65+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Susana Miguel, MSc, MD, PhD candidate, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025.08868.SAU+
Record Dates: First submitted 2025-11-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight; Aged 65 Years or Older
Keywords: Aged; Overweight; Snack exercise; Community Health Planning
MeSH Terms: conditions — Obesity; Overweight | interventions — Prescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief educational counselling session (Active Comparator): Participants will receive a brief educational counselling session (60 minutes) at the baseline assessment. This session will be a standardized brief educational counseling session delivered by trained research personnel during the baseline assessment. This session will provide foundational information on the benefits of physical activity for healthy aging and offer practical strategies for incorporating short "physical activity snacks" into daily routines. This ensures a consistent educational baseline for both study arms.
  Interventions: Behavioral: Brief educational counseling session
- Brief educational counselling session + Group-based "Snack Exercise" training and prescription (Active Comparator): Participants will receive a standardized Brief Educational Counselling Session at baseline. This group will then proceed with the Structured Community-based Physical Activity Snack Intervention (COMPASS 65+). The program will consist of group-based, theory-based and practical sessions (held 2-3 times per week, each lasting approximately 45 minutes).
  Interventions: Behavioral: Group-based "Snack Exercise" Training and Prescription; Behavioral: Brief educational counseling session

INTERVENTIONS:
Behavioral: Group-based "Snack Exercise" Training and Prescription — This programme consists of supervised, group-based sessions (2-3 per week, ~45 minutes each) combining concise theoretical instruction with guided practical execution of the snack-exercise protocol. Sessions are delivered by a qualified exercise professional and focus on teaching correct technique, safety, and progression of the prescribed short exercise bouts ("exercise snacks").
  At the end of each session, participants receive an individualized home-based exercise prescription, tailored to their functional capacity and progression markers. Exercise intensity during supervised and home practice is monitored using the OMNI-BORG perceived exertion scale, progressing from light to moderate intensity, in accordance with World Health Organization recommendations.
  Arms: Brief educational counselling session + Group-based "Snack Exercise" training and prescription
Behavioral: Brief educational counseling session — A standardized brief educational counseling session delivered by trained research personnel during the baseline assessment. This session will provide foundational information on the benefits of physical activity for healthy aging and offer practical strategies for incorporating short "physical activity snacks" into daily routines. This ensures a consistent educational baseline for both study arms.

SUMMARY:
This study will explore a new way for older adults to become more physically active. As people get older, it's common to gain weight and lose muscle strength. This combination can make it harder to do daily activities, increase the risk of falls, and impact overall quality of life. While we know that regular exercise is very beneficial, many older adults find it difficult to stick to traditional exercise programs due to lack of time, motivation, or energy.

This research project, called COMPASS 65+, will test an innovative approach called "snack exercise." Instead of one long workout, "snack exercise" involves doing several short bouts of activity, a few minutes at a time, throughout the day. The main idea is that these short, frequent bouts of activity might be easier to fit into a daily routine and less tiring than longer exercise sessions.

The purpose of this study is to see if a "snack exercise" program is a feasible and enjoyable way for adults aged 65 and over, who are overweight or obese, to improve their health. The study will be conducted in two main parts. First, the research team will talk with older adults to understand what helps or hinders them from being active to co-design the program. Second, volunteers will be randomly assigned to either a "snack exercise" group or a control group.

Participants in the "snack exercise" group will attend sessions that combine theory and practice to learn how to perform these exercises and will receive individualized prescriptions to perform the "snacks" (short bouts) at home. The control group will receive a brief educational counselling session on physical activity. Participants' health status, body composition, and physical fitness will be assessed at baseline, after the 12 weeks intervention, and again 6 weeks post-intervention to evaluate the maintenance of any improvements. These outcomes will help determine whether short bouts of 'exercise snacking' constitute a feasible and effective strategy to promote functional capacity, metabolic health, and long-term adherence to physical activity.

DETAILED DESCRIPTION:
Study Rationale and Background The intersection of an aging population and the obesity epidemic poses a significant public health challenge, particularly for adults aged 65 and older. This combination often leads to sarcopenic obesity, a condition characterized by excess body fat and low muscle mass and strength, which substantially increases the risk of falls, frailty, functional decline, and loss of independence. While physical activity is a proven non-pharmacological intervention to counteract these declines, adherence to traditional, structured exercise programs remains low among older adults. Barriers such as a perceived lack of time, low motivation, and fatigue create a gap between the known benefits of exercise and its practical implementation in real-world community settings.

This study, COMPASS 65+, proposes to evaluate an innovative exercise modality known as "snack exercise." This approach involves short, frequent bouts of physical activity performed throughout the day, designed to be more accessible and less burdensome than conventional exercise routines. The primary aim of this project is to assess the feasibility, acceptability, and preliminary effects of a community-based "snack exercise" program, co-designed with input from the target population, for overweight and obese older adults. The findings are intended to provide the necessary evidence to design a future, definitive large-scale randomized controlled trial (RCT).

Study Design

The research plan is structured in two sequential phases:

1. Phase 1: Exploratory Mixed-Methods Study This initial phase is designed to inform the development of the intervention. It involves a mixed-methods approach to identify barriers, facilitators, and preferences related to physical activity among the target population.

   * Quantitative Component: A cross-sectional survey will be administered to a convenience sample of 370 adults aged 65 or older with a Body Mass Index (BMI) of 25 kg/m² or greater. The survey will include validated instruments such as the Exercise Benefits/Barriers Scale (EBBS) and the Multimorbidity Treatment Burden Questionnaire (MTBQ).
   * Qualitative Component: Focus groups will be conducted with a randomly selected subset of the target population to explore user preferences for program design.The data will be integrated to co-design a "snack exercise" intervention that is evidence-based and tailored to user needs.
2. Phase 2: Feasibility Randomized Controlled Trial (RCT) A two-arm, parallel-group feasibility RCT will be conducted to test the co-designed intervention.

   * Participants: A target of 60 participants will be recruited from primary care settings. Inclusion criteria include adults aged ≥ 65 years with a BMI ≥ 25 kg/m². Exclusion criteria include significant cognitive deficits, contraindications to exercise (assessed via PAR-Q+), major cardiovascular events within the last 3 months, unstable chronic disease, or severe mobility impairment.
   * Randomization: Participants will be randomly allocated (1:1) to either the intervention group or the control group.
   * Timeline: The intervention lasts 12 weeks, followed by a 6-week post-intervention "washout" period. Assessments occur at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
   * Intervention Groups Active Comparator (Control Group): Participants will receive a single, standardized Brief Educational Counselling Session (60 minutes) at baseline (T0). Delivered by trained research personnel, this session provides foundational information on the benefits of physical activity for healthy aging and offers practical strategies for incorporating short "physical activity snacks" into daily routines. This ensures a consistent educational baseline.

Experimental Group ("Snack Exercise"): Participants will receive the standardized Brief Educational Counselling Session at baseline, followed by the Structured Community-based Physical Activity Snack Intervention. This program consists of group-based, theoretico-practical sessions held 2-3 times per week, each lasting approximately 45 minutes. Sessions are guided by a physical exercise professional and focus on explaining and practicing the prescribed snack exercises. Crucially, at the end of each session, participants are provided with an individualized physical prescription to perform at home. Exercise intensity is monitored using perceived exertion scales (BORG-OMNI), progressing from light to moderate intensity per WHO recommendations.

Study Procedures and Outcome Measures Protocol & Ethics: The study adheres to SPIRIT guidelines and the Declaration of Helsinki, with Ethics Committee approval and written informed consent required.

Outcomes & Data Collection: Comprehensive assessments are conducted at T0, T1, and T2 using validated instruments and objective tools:

* Body Composition & Anthropometrics: Dual-Energy X-ray Absorptiometry (DEXA) for fat/lean mass and bone density; Height, Weight, BMI (kg/m^2), and Waist Circumference.
* Cardiorespiratory Fitness: One-Mile Walk Test to predict aerobic capacity (VO2 max).
* Functional Fitness & Fall Risk: The Short Physical Performance Battery (SPPB) (assessing balance, gait speed, and chair stands) and the 30-second Chair Stand Test (muscular endurance).
* Stability: Limits of stability assessed via a force platform (Physiosensing®).
* Daily Physical Activity: Objectively measured using a Fitband worn for five consecutive days (step count, active minutes).
* Psychosocial & Health Status: Exercise Self-Efficacy Scale (ESES).
* Multidimensional Lifestyle and Health Status (assessed via the Healthy Lifestyle Assessment Toolkit, covering cardiometabolic health, well-being, nutrition, mental health, and sleep).

Statistical Analysis Plan Primary Analysis (Feasibility): Descriptive analysis of recruitment, adherence, retention, and protocol fidelity based on the RE-AIM framework.

Secondary Analysis (Preliminary Effects): Repeated measures ANOVA or mixed models will be used to assess changes over time (T0, T1, T2) and between groups (p< 0.05). The goal is to estimate effect sizes to power a future definitive trial.

Data Management: All analyses will be conducted using SPSS (Version 29), with appropriate handling of missing data (e.g., multiple imputation).

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≥65 years with a BMI ≥25 kg/m².

Exclusion Criteria:

* significant cognitive deficits,
* contraindications to exercise (assessed via PAR-Q+),
* major cardiovascular events within the last 3 months,
* unstable chronic disease,
* severe mobility impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (Reach) | From the start of recruitment until the target sample size is reached (approximately 2 months).
  The percentage of eligible individuals who consent to participate in the study out of all individuals invited. This will be a measure of the reach and appeal of the intervention and study design.
Adherence to the "Snack Exercise" Program (Effectiveness) | Throughout the 12-week intervention period.
  The percentage of scheduled "snack exercise" sessions attended by participants in the intervention group. Adherence will be calculated as (number of sessions attended / total number of scheduled sessions) x 100. This measures the effectiveness of the program in engaging participants.
Program Implementation Fidelity (Implementation) | Throughout the 12-week intervention period.
  The degree to which the "snack exercise" program is delivered as intended by the study protocol. This will be assessed by a checklist monitoring staff adherence to the protocol, including session content, duration, and intensity monitoring procedures. It will be measured as a percentage of protocol items successfully delivered.
Participant Retention Rate | From baseline (T0) to the final follow-up assessment (T2) at 18 weeks.
  The percentage of enrolled participants who complete all study assessments at all time points (T0, T1, and T2). This measures the overall acceptability of the study procedures and the ability to retain participants over the full duration.
Intention to Continue Exercise (Maintenance) | At the final follow-up assessment (T2) at 18 weeks.
  Assessed via a self-report questionnaire administered at the final follow-up visit, evaluating participants' intention and confidence to continue with "snack exercise" or other forms of physical activity independently after the study concludes.

SECONDARY OUTCOMES:
Multidimensional Lifestyle and Health Status | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Evaluated using the Healthy Lifestyle Assessment Toolkit, a comprehensive instrument that assesses multiple domains including cardiometabolic health (blood pressure), well-being, nutrition, mental health, sleep quality, and self-perceived health status. The toolkit identify risks and guide interventions, using systems like traffic light scores (green/yellow/orange) for feedback and promoting behavior change for better health outcomes.
Daily Physical Activity Patterns | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Objectively measured using a triaxial accelerometer (worn on the hip for 5-7 consecutive days). Participants will be instructed to wear the device during all waking hours, removing it only for water-based activities or sleeping. The accelerometers provided objective measures of daily movement patterns, including step count, time spent in different activity intensities, and sedentary behavior. This approach allow us to evaluate changes in physical activity levels throughout the intervention and to assess adherence.
Body Composition - Dual-Energy X-ray Absorptiometry (DEXA) | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Assessed using Dual-Energy X-ray Absorptiometry (DEXA) to measure changes in fat mass, lean mass, and bone mineral density.
Anthropometrics - Height | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Anthropometric measures including height - height in meters (m).
Anthropometrics - Weight | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Anthropometric measures including Weight - weight in kilograms (kg).
Anthropometrics - Body Mass Index (BMI) | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Anthropometric measures including Body Mass Index (BMI) - weight in kilograms by height in meters squared (kg/m^2).
Anthropometrics - Waist circumference | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Anthropometric measures including waist circumference will also be collected - waist circumference in cm.
Cardiorespiratory Fitness | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Assessed using the One-Mile Walk Test (1,61 kilometers) for evaluation of cardiovascular fitness, to predict an individual's aerobic capacity, also known as maximal oxygen consumption (VO2 max).
  A slower time indicates lower cardiorespiratory fitness, and it's also a strong predictor of health outcomes.
Functional Fitness (muscular endurance) | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  A battery of tests will be used, including the 30-second chair stand test for muscular endurance. This measures lower body muscular endurance by counting how many times a person can stand up from a chair and sit back down in 30 seconds, using arms folded across the chest for support.
  Scores decline with age. A below average score (in seconds) indicates a risk for falls, being the cut off for each age group:
  65-69: < 12 (M); < 11 (W) 70-74: < 12 (M); < 10 (W) 75-79: < 11 (M); < 10 (W) 80-84: < 10 (M); < 9 (W) 85-89: < 8 (M); < 8 (W) 90-94: < 7 (M); < 4 (W)
Functional Fitness and Fall risk - Short Physical Performance Battery (SPPB) | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  A battery of tests will be used, including the Short Physical Performance Battery (SPPB) for functional capacity and fall risk. This is an objective test for older adults assessing lower-body function via 3 tasks: standing balance, usual gait speed (4m walk), and chair stands (5 reps, arms crossed). Scoring 0-12 (higher is better), predict disability, falls, hospitalization, and mortality, and is highly reliable for measuring physical capability in various settings.
Fall Risk and Functional stability (force platform) | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Assessment of limits of stability using a force platform for functional stability (Physiosensing® v.19002, Sensing Future, Coimbra, Portugal).
Exercise Self-Efficacy (ESES) | Assessed at baseline (T0), post-intervention (T1, 12 weeks), and follow-up (T2, 18 weeks).
  Assessed using the Exercise Self-Efficacy Scale (ESES), a self-report measure to evaluate participants' confidence in their ability to engage in exercise. Participants answer on a 4-point rating scale, possible scoring range 10-40. A higher total score means greater exercise self-efficacy (stronger belief in one's ability to exercise).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos S Cardoso, PhD, MD, Study Director — University of Coimbra; Anabela M Pinto, PhD, MD, Study Chair — University of Coimbra; Susana P Miguel, MSc, MD, Principal Investigator — University of Coimbra; Guilherme Eustáquio Furtado, PhD, Study Chair — Polytechnic Institute of Coimbra
Locations (1):
- Fernão de Magalhães Health Center, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
A plan for sharing individual participant data with external researchers has not been established at this stage for several reasons. Primarily, this is a feasibility study with a small sample size, designed to inform the design of a future, larger trial rather than to produce generalizable findings. Due to the small cohort and specific regional recruitment, there is a potential risk of deductive disclosure of participant identity, even with de-identified data. Furthermore, the informed consent obtained from participants does not include a specific clause for sharing their individual data beyond the core research team for secondary research purposes. Therefore, to uphold ethical commitments to participant confidentiality, IPD will not be made available at the conclusion of this study.

REFERENCES:
- [Background] Reis F, Sa-Moura B, Guardado D, Couceiro P, Catarino L, Mota-Pinto A, Verissimo MT, Teixeira AM, Ferreira PL, Lima MP, Palavra F, Rama L, Santos L, van der Heijden RA, Goncalves CE, Cunha A, Malva JO. Development of a Healthy Lifestyle Assessment Toolkit for the General Public. Front Med (Lausanne). 2019 Jun 27;6:134. doi: 10.3389/fmed.2019.00134. eCollection 2019. PMID 31316985
- [Background] Vancea A, Iliescu M, Aivaz KA, Popescu MN, Beiu C, Spiru L. Improving Functional Capacities and Well-Being in Older Adults: Strategies in Physical Medicine and Rehabilitation. Cureus. 2024 Aug 6;16(8):e66254. doi: 10.7759/cureus.66254. eCollection 2024 Aug. PMID 39238764
- [Background] Rodrigues RN, Carballeira E, Silva F, Caldo-Silva A, Abreu C, Furtado GE, Teixeira AM. The Effect of a Resistance Training, Detraining and Retraining Cycle on Postural Stability and Estimated Fall Risk in Institutionalized Older Persons: A 40-Week Intervention. Healthcare (Basel). 2022 Apr 22;10(5):776. doi: 10.3390/healthcare10050776. PMID 35627913
- [Background] Nuzzo JL, Pinto MD, Kirk BJC, Nosaka K. Resistance Exercise Minimal Dose Strategies for Increasing Muscle Strength in the General Population: an Overview. Sports Med. 2024 May;54(5):1139-1162. doi: 10.1007/s40279-024-02009-0. Epub 2024 Mar 20. PMID 38509414
- [Background] Lee PG, Jackson EA, Richardson CR. Exercise Prescriptions in Older Adults. Am Fam Physician. 2017 Apr 1;95(7):425-432. PMID 28409595
- [Background] Hashimoto K, Dora K, Murakami Y, Matsumura T, Yuuki IW, Yang S, Hashimoto T. Positive impact of a 10-min walk immediately after glucose intake on postprandial glucose levels. Sci Rep. 2025 Jul 2;15(1):22662. doi: 10.1038/s41598-025-07312-y. PMID 40594496
- [Background] Evans K, Abdelhafiz D, Abdelhafiz AH. Sarcopenic obesity as a determinant of cardiovascular disease risk in older people: a systematic review. Postgrad Med. 2021 Nov;133(8):831-842. doi: 10.1080/00325481.2021.1942934. Epub 2021 Jul 12. PMID 34126036
- [Background] Eitmann S, Matrai P, Hegyi P, Balasko M, Eross B, Dorogi K, Petervari E. Obesity paradox in older sarcopenic adults - a delay in aging: A systematic review and meta-analysis. Ageing Res Rev. 2024 Jan;93:102164. doi: 10.1016/j.arr.2023.102164. Epub 2023 Dec 14. PMID 38103840
- [Background] Collado-Mateo D, Lavin-Perez AM, Penacoba C, Del Coso J, Leyton-Roman M, Luque-Casado A, Gasque P, Fernandez-Del-Olmo MA, Amado-Alonso D. Key Factors Associated with Adherence to Physical Exercise in Patients with Chronic Diseases and Older Adults: An Umbrella Review. Int J Environ Res Public Health. 2021 Feb 19;18(4):2023. doi: 10.3390/ijerph18042023. PMID 33669679
- [Background] Campisi J, Kapahi P, Lithgow GJ, Melov S, Newman JC, Verdin E. From discoveries in ageing research to therapeutics for healthy ageing. Nature. 2019 Jul;571(7764):183-192. doi: 10.1038/s41586-019-1365-2. Epub 2019 Jul 10. PMID 31292558